CLINICAL TRIAL: NCT03142373
Title: Variations of Heart Rate Variability and Skin Conductance Reveal the Influence of CV4 and Rib Raising Osteopathic Techniques on the Autonomic Nervous System: a Randomized Controlled Trial
Brief Title: Effect of CV4 and Rib Raising Techniques on Autonomic Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Chiara Arienti, Dr, Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OMT and HRV
Record Dates: First submitted 2017-04-28; First posted 2017-05-05 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Autonomic Nervous System Disease; Osteopathy
Keywords: heart rate variability; autonomic nervous system; osteopathic manipulative treatment; skin conductance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CV4 group (Experimental): CV4 technique
  Interventions: Other: CV4 technique
- RR group (Experimental): Rib Raising technique
  Interventions: Other: RR technique
- Placebo group (Placebo Comparator): Light touch
  Interventions: Other: Placebo treatment

INTERVENTIONS:
Other: CV4 technique
  Arms: CV4 group
Other: RR technique
  Arms: RR group
Other: Placebo treatment
  Arms: Placebo group

SUMMARY:
Background. Heart rate variability (HRV) and skin conductance (SC) highlight autonomic activity and the balance of autonomic nervous system (ANS) which regulates involuntary physiological functions. The modulation of ANS tonic activity is a target of osteopathic manipulative treatment (OMT). The main aim of the present study was to verify whether CV4 and RR osteopathic techniques influence ANS activity.

Trial design. A randomized-controlled clinical trial was performed from June 2010 to January 2011.

Methods. 32 healthy adults were selected. At enrollment, all healthy subjects were randomized in three groups: CV4 group (CV4 technique), Rib Raising group (RR technique), and Placebo group (PL technique). HRV and SC was recorded during the session respectively with heart rate monitor Polar S810i and with Onda Scanner Domiana (OSD-Microsale model). All data analysis was performed using SPSS statistical software and the significance level set at p≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* between 18-65 years old
* both gender

Exclusion Criteria:

* BMI ≥ 30
* pregnancy
* menstrual flow during the session
* chronic pain
* chronic drug treatment
* presence of skin, cardiovascular, psychiatric and neurological diseases
* medical history of surgical interventions
* OMT in the previous 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | 1200 seconds
  HRV was measured using a heart rate monitor Polar S810i frequency meter

SECONDARY OUTCOMES:
Skin Conductance | 1200 seconds
  SC was measured using a Onda Scanner Domiana (OSD-Microsale model).

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Arienti, PhD, Principal Investigator — IRCCS Don Gnocchi Foundation

IPD SHARING:
Plan to Share IPD: Undecided